CLINICAL TRIAL: NCT01565902
Title: A Single-dose, Open-label, Parallel-group Study to Assess the Pharmacokinetics of BAF312 in Subjects With Mild, Moderate and Severe Hepatic Impairment Compared to Healthy Control Subjects.
Brief Title: Pharmacokinetics of BAF312 in Patients With Hepatic Impairment
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: CBAF312A2122; 2012-000562-37 (EudraCT Number)
Record Dates: First submitted 2012-03-26; First posted 2012-03-29 (Estimated); Results first posted 2014-12-22 (Estimated); Last update posted 2020-12-29 (Actual); Status verified 2018-02

CONDITIONS: Hepatic Impairment
Keywords: BAF312; Pharmacokinetics; Hepatic impairment
MeSH Terms: interventions — siponimod

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- Mild hepatically impaired (Experimental): Treatment with a single oral dose of 0.25 mg BAF312
  Interventions: Drug: BAF312
- Moderate hepatically impaired (Experimental): Treatment with a single oral dose of 0.25 mg BAF312
  Interventions: Drug: BAF312
- Severe hepatically impaired (Experimental): Treatment with a single oral dose of 0.25 mg BAF312
  Interventions: Drug: BAF312
- Matched healthy subjects (Experimental): Treatment with a single oral dose of 0.25 mg BAF312
  Interventions: Drug: BAF312

INTERVENTIONS:
Drug: BAF312 — Treatment with a single oral dose of 0.25 mg BAF312

SUMMARY:
This study will investigate the pharmacokinetics of BAF312 in patients with mild, moderate and severe hepatic impairment compared to healthy control subjects.

ELIGIBILITY:
Inclusion Criteria:

All subjects:

* Male and female Caucasian subjects 18 to 70 years of age
* At least 50 kg and body mass index (BMI) within 18-35 kg/m2.
* CYP2C9 wild-type (CYP2C9*1 homozygous carriers)

Hepatic impairment:

- Subjects must have either mild, moderate or severe hepatic impairment

Exclusion Criteria:

All subjects

* Hepatic impairment due to non-liver disease.
* Use of other investigational drugs within certain timelines
* Donation or loss of 400 mL or more of blood or plasma within eight (8) weeks prior to initial dosing
* History of cardiac rhythm abnormalities or cardiac rhythm abnormalities identified in the 24-h Holter ECG recording including episodes of bradycardia (HR < 50 bpm) during waking hours and/or arrhythmic episodes; subjects with history or presence of ventricular rhythm disturbances (ventricular extra-systoles >100/24h, or higher grade), or supraventricular arrhythmias (other than occasional supraventricular ectopic beats with a maximum of 5 subsequent ectopic beats per event) or subjects with conduction disturbances (higher than AV-block grade 1) or bradycardia or tachycardia.
* History of cardiac catheter ablation.
* Women of child-bearing potential
* History of malignancy of any organ system
* Recent and/or recurrent history of acute or chronic bronchospastic disease (including asthma and chronic obstructive pulmonary disease)
* History or presence of symptomatic postural hypotension or syncope.
* Total WBC or lymphocyte counts which falls outside the 1.5-fold local laboratory normal range or platelet count < 30,000/μL at screening or baseline.
* Clinically significant infection or recent vaccination with live-attenuated vaccines.
* History or presence of hepatitis B or C and/or positive Hepatitis B surface antigen (HBsAg) or Hepatitis C test result at screening.
* History or presence of coronary heart disease (stable or unstable), myocardial infarction, myocarditis, cardiomyopathy, heart failure NYHA II - IV.

Hepatic impairment:

* History or presence of any non-controlled and clinically significant disease that could affect the study outcome or that would place the patient at undue risk.
* Any surgical or medical condition other than hepatic impairment which might significantly alter the absorption, distribution, metabolism, or excretion of drugs, or which may jeopardize the safety of the study subject in case of participation in the study.
* Treatment with certain drugs

Healthy subjects:

* History or presence of any clinically significant disease of any major system organ class including (but not limited to) cardiovascular, metabolic, renal, neurological or psychiatric diseases.
* Any surgical or medical condition which might significantly alter the absorption, distribution, metabolism, or excretion of drugs, drugs, or which may jeopardize the subject in case of participation in the study.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2012-10; Primary Completion 2014-03 (Actual); Study Completion 2014-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (3):
- Hungary (2):
  - Novartis Investigative Site, Balatonfüred
  - Novartis Investigative Site, Budapest
- Novartis Investigative Site, Moscow, Russia

REFERENCES:
- See also: Publication from the International Journal of Clinical Pharmacology and Therapeutics — https://www.dustri.com/nc/article-response-page.html?artId=14609&doi=10.5414%2FCP202588
- See also: Results for CBAF312A2122 can be found on the Novartis Clinical Trial Results Website — https://www.novctrd.com/ctrdweb/trialresult/trialresults/pdf?trialResultId=13203

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Up to forty-eight subjects were planned to be enrolled in four groups. A total of 40 subjects were enrolled and completed the study. All subjects were included in the safety and PK analysis. However, only 38 subjects were included for primary PK analysis based on matched pair analysis
Pre-assignment Details: To potentially reduce the number of healthy subjects exposed to BAF312, study allowed for multiple matching of subjects with hepatic impairment to healthy subjects. During the study, 2 healthy subjects were not matched to any of the subjects with hepatic impairment due to a retrospective identification of a better matching partner
Period: Overall Study
Arm/Group | Mild Hepatically Impaired | Moderate Hepatically Impaired | Severe Hepatically Impaired | Matched Healthy Subjects
Started | 8 | 8 | 8 | 16
Completed | 8 | 8 | 8 | 16
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Mild Hepatically Impaired | Moderate Hepatically Impaired | Severe Hepatically Impaired | Matched Healthy Subjects | Total
Number analyzed (Participants) | 8 | 8 | 8 | 16 | 40
Age, Continuous [Mean (Standard Deviation); unit: Years] | 53.9 (6.20) | 47.8 (6.30) | 51.8 (3.41) | 50.1 (5.50) | 50.7 (5.65)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 2 | 4 | 6 | 14
  Male | 6 | 6 | 4 | 10 | 26

OUTCOME MEASURES:

1. Primary Outcome: Pharmacokinetic Parameters of BAF312 and Selected Metabolites: Area Under the Plasma Concentration-time Curve From Time Zero to Infinity (AUCinf)
Description: The pharmacokinetics of BAF312 were studied in plasma up to 504 hours post-dose at the following time points: pre-dose, 0.25, 0.5, 0.75, 1, 1.5, 2, 3, 4, 6, 8, 12, 16, 24, 36, 48, 72, 96, 144, 216, 312, 408 and 504 hours post dose.
Time Frame: pre-dose, 0.25, 0.5, 0.75, 1, 1.5, 2, 3, 4, 6, 8, 12, 16, 24, 36, 48, 72, 96, 144, 216, 312, 408 and 504 hours post dose.
Population: The PK analysis set consists of all completed subjects with quantifiable pharmacokinetic (PK) measurements. To reduce the number of healthy subjects exposed to BAF312, study allowed matching of subjects with hepatic impairment to healthy subjects. A healthy subject served as matching partner for up to 3 subjects with hepatic impairment
Measure: Mean (Standard Deviation); unit: h*ng/mL
Groups:
- Matched Healthy Subjects - Mild; Matched Healthy Subjects - Moderate; Matched Healthy Subjects - Severe: Treatment with a single oral dose of 0.25 mg BAF312
Arm/Group | Mild Hepatically Impaired | Moderate Hepatically Impaired | Severe Hepatically Impaired | Matched Healthy Subjects - Mild | Matched Healthy Subjects - Moderate | Matched Healthy Subjects - Severe
Number analyzed (Participants) | 8 | 7 | 8 | 8 | 8 | 8
h*ng/mL | 68.3 (24.5) | 53.9 (7.57) | 73.7 (25.4) | 64.2 (20.8) | 63.2 (18.6) | 64.9 (23.6)

2. Primary Outcome: Pharmacokinetic Parameters of BAF312 and Selected Metabolites: Area Under the Plasma Concentration-time Curve From Time Zero to the Time of the Last Quantifiable Concentration (AUClast)
Description: as for outcome 1
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: h*ng/mL
Arm/Group | Mild Hepatically Impaired | Moderate Hepatically Impaired | Severe Hepatically Impaired | Matched Healthy Subjects - Mild | Matched Healthy Subjects - Moderate | Matched Healthy Subjects - Severe
Number analyzed (Participants) | 8 | 7 | 8 | 8 | 8 | 8
h*ng/mL | 66.8 (24.4) | 52.3 (7.51) | 71.6 (24.5) | 62.5 (20.9) | 61.7 (18.7) | 63.4 (23.6)

3. Primary Outcome: Pharmacokinetic Parameters of BAF312 and Selected Metabolites: Observed Maximum Plasma Concentration Following Drug Administration at Steady State (Cmax)
Description: as for outcome 1
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: (ng/mL)
Arm/Group | Mild Hepatically Impaired | Moderate Hepatically Impaired | Severe Hepatically Impaired | Matched Healthy Subjects - Mild | Matched Healthy Subjects - Moderate | Matched Healthy Subjects - Severe
Number analyzed (Participants) | 8 | 7 | 8 | 8 | 8 | 8
(ng/mL) | 2.03 (0.532) | 1.54 (0.191) | 1.58 (0.304) | 1.74 (0.439) | 1.80 (0.417) | 1.94 (0.603)

4. Secondary Outcome: Number of Patients With Adverse Events, Serious Adverse Events and Death Adverse Events (Frequency of Adverse Events, Serious Adverse Events, and Notable Laboratory Abnormalities) of of BAF312 After a Single Dose of BAF312
Description: Physical examination, vital signs, body temperature, standard safety laboratory evaluations (hematology, clinical chemistry, coagulation, Hepatitis B and C and HIV serology, α-fetoprotein [in hepatically impaired subjects only], pregnancy test, alcohol and drug screen), standard 12-lead electrocardiogram , cardiac monitoring, 24-h Holter ECG, suicidality assessment (C-SSRS), (serious) adverse event monitoring.
Time Frame: Day -1 to 22
Population: The safety analysis set consists of all subjects that received study drug and with no protocol deviations with relevant impact on safety.
Measure: Number; unit: Participants
Arm/Group | Mild Hepatically Impaired | Moderate Hepatically Impaired | Severe Hepatically Impaired | Matched Healthy Subjects
Number analyzed (Participants) | 8 | 8 | 8 | 16
Participants
  At least one AE | 0 | 1 | 1 | 1
  Serious Adverse Events | 0 | 0 | 0 | 0
  Death | 0 | 0 | 0 | 0

ADVERSE EVENTS:
Arm/Group | Moderate Hepatically Impaired | Severe Hepatically Impaired | Matched Healthy Subjects | Mild Hepatically Impaired
Serious Adverse Events (participants affected / at risk) | 0/8 | 0/8 | 0/16 | 0/8
Other Adverse Events (participants affected / at risk) | 1/8 | 1/8 | 1/16 | 0/8
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Moderate Hepatically Impaired (N=8) | Severe Hepatically Impaired (N=8) | Matched Healthy Subjects (N=16) | Mild Hepatically Impaired (N=8)
Atrioventricular block first degree (Cardiac disorders) | 0 | 1 | 0 | 0
Tonsillitis (Infections and infestations) | 1 | 0 | 0 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (i.e., data from all sites) in the clinical trial or disclosure of trial results in their entirety